CLINICAL TRIAL: NCT00514826
Title: Study to Investigate Sleep Apnea Patients at Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Konrad E. Bloch, Professor, MD, University Hospital of Zurich, Switzerland
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: EK1413
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: altitude exposure — sojourn at moderate altitude (1860m and 2590m) during 2 days/nights each

SUMMARY:
The purpose of the study is to investigate the effect of an altitude sojourn on patients with the obstructive sleep apnea syndrome

DETAILED DESCRIPTION:
Previous observations do not allow to draw firm conclusions on the effect of altitude sojourn on sleep, breathing and daytime performance in patients with the obstructive sleep apnea syndrome. Furthermore, the susceptibility of sleep apnea patients to high altitude related illness is not known. Therefore, the purpose is to study untreated patients with obstructive sleep apnea syndrome living at low altitude during a sojourn of a few days at moderate altitude in order to evaluate the physiologic effects of hypobaric hypoxia in these patients. We hypothesize that: 1. Sleep and nocturnal breathing disturbances in untreated OSA patients are more pronounced at moderate altitude compared to low altitude. 2. The increase in sleep related breathing disturbances at moderate altitude is due to an increase in central apnea/hypopnea

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnea syndrome based on symptoms and a sleep study

Exclusion Criteria:

* Sleep disorders other than obstructive sleep apnea syndrome
* Other than mild, stable cardiovascular disease
* Other than mild lung disease
* Chronic rhinitis, previous uvulopalatopharyngoplasty
* Treatment with drugs that affect respiratory center drive
* Internal, neurologic or psychiatric disease that interferes with sleep quality
* Previous intolerance to moderate or low altitude < 2600m

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Prevalence and severity of sleep disordered breathing | during altitude sojourn

SECONDARY OUTCOMES:
alterations in sleep structure and vigilance; high altitude related illness | during altitude sojourn

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E. Bloch, MD, Study Director — Pulmonary Division, University Hospital Zurich, Switzerland
Locations (1):
- Pulmonary Division, University Hospital Zurich, Switzerland, Zurich, Switzerland

REFERENCES:
- [Result] Nussbaumer-Ochsner Y, Schuepfer N, Ulrich S, Bloch KE. Exacerbation of sleep apnoea by frequent central events in patients with the obstructive sleep apnoea syndrome at altitude: a randomised trial. Thorax. 2010 May;65(5):429-35. doi: 10.1136/thx.2009.125849. PMID 20435865
- [Derived] Bloch KE, Latshang TD, Turk AJ, Hess T, Hefti U, Merz TM, Bosch MM, Barthelmes D, Hefti JP, Maggiorini M, Schoch OD. Nocturnal periodic breathing during acclimatization at very high altitude at Mount Muztagh Ata (7,546 m). Am J Respir Crit Care Med. 2010 Aug 15;182(4):562-8. doi: 10.1164/rccm.200911-1694OC. Epub 2010 May 4. PMID 20442435